CLINICAL TRIAL: NCT04366245
Title: Phase I / II Multicentre, Randomized and Controlled Clinical Trial to Evaluate the Efficacy of Treatment With Hyperimmune Plasma Obtained From Convalescent Antibodies of COVID-19 Infection
Brief Title: Clinical Trial to Evaluate the Efficacy of Treatment With Hyperimmune Plasma Obtained From Convalescent Antibodies of COVID-19 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC/COVID-19
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV 2
MeSH Terms: interventions — COVID-19 Serotherapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Biological: Hyperimmune plasma
- Comparator (Active Comparator)
  Interventions: Drug: Standard of care for SARS-CoV-2 infection

INTERVENTIONS:
Biological: Hyperimmune plasma — PLASMA OF CONVALESCENT COVID-19
  Arms: Experimental
Drug: Standard of care for SARS-CoV-2 infection — Standard of care for SARS-CoV-2 infection
  Arms: Comparator

SUMMARY:
Phase I / II multicentre, randomized and controlled clinical trial to evaluate the efficacy of treatment with hyperimmune plasma obtained from convalescent antibodies of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent prior to performing procedures. the oral consent be accepted testified to prevent paper handling.
2. Patient of both sexes, and ≥18 years.
3. SARS-CoV-2 infection determined by PCR in a sample of naso-oropharyngeal exudate or other respiratory specimen or determination of specific positive IgM antibodies, in <72 hours before randomization.
4. Patients requiring hospitalization for pneumonia COVID-19 without need until randomization of mechanical ventilation (invasive or non-invasive), and at least one of the following:

   * O2 saturation ≤ 94% in ambient air, or PaO2 / FiO2 ≤ 300 mm Hg.
   * Age> 65 years.
   * Presence of: high blood pressure, chronic heart failure, chronic obstructive pulmonary disease, liver cirrhosis, or other chronic pulmonary and cardiovascular diseases, diabetes, or obesity

Exclusion Criteria:

1. Requirement before randomization of mechanical ventilation (invasive or non-invasive).
2. Any of the following analytical data before randomization: IL-6> 80 pg / mL, D-dimer> 10 times ULN, ferritin> 1000ng / mL.
3. Participation in another clinical trial or experimental treatment for COVID-19.
4. In the opinion of the clinical team, progression to death or mechanical ventilation is highly probable within 24 hours, regardless of treatment provision.
5. Incompatibility or allergy to the administration of human plasma.
6. Severe chronic kidney disease grade 4 or requiring dialysis (ie eGFR <30)
7. Pregnant, lactating, or fertile women who are not using an effective method of contraception. It is considered a woman of childbearing age all women from 18 years and up to a year after the last menstrual period in the case of menopausal women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of Adverse Events and Serious Adverse Events grade 3 and 4, related to the product under investigation or the administration procedure, graduated according to the common toxicity criteria scale (CTCAE). | 30 days after enrollment
  Incidence of Adverse Events and Serious Adverse Events grade 3 and 4, related to the product under investigation or the administration procedure, graduated according to the common toxicity criteria scale (CTCAE).
Efficacy: Death from any cause | Day +21 after randomization
Efficacy: Need for mechanical ventilation | Day +21 after randomization
Efficacy: Any of the following analytical data after 72h of randomization. | Day +21 after randomization
  IL-6> 80 pg / mL, D-dimer> 10 times, ferritin> 1000 ng / mL.
Efficacy: SOFA scale ≥ 3 after 72 hours of randomization or an increase of 2 points or more from the basal level | Day +21 after randomization

SECONDARY OUTCOMES:
Efficacy. Mortality on days 14 and 28. | Days 14 and 28.
Efficacy: Proportion of patients who required mechanical ventilation | Until day 28
Efficacy: Proportion of patients who develop analytical alterations. | Day +21 after randomization.
  IL-6> 80 pg / mL, D-dimer> 10 times, ferritin> 1000 ng / mL until the cure test.
Efficacy: Cure / clinical improvement (disappearance or improvement of signs and symptoms of COVID-19) in the cure test. | Day +21 after randomization
Efficacy: PCR negative for SARS-CoV-2 | On days 7 and 21
Efficacy: Proportion of patients requiring treatment. | Until day 21.
  Proportion of patients requiring treatment with Tocilizumab Sarilumab, Anakimra or other IL-6 or IL-1 antagonists, or corticosteroids at doses of methylprednisolone greater than 2 mg / Kg / day (or equivalent) and / or any investigational medication.
Efficacy: Duration of hospitalization (days) | Until day 21.
Virology and immunological variables: Qualitative PCR for SARS-CoV-2 in naso-oropharyngeal exudate sample | At baseline and on day 21
Virology and immunological variables: Total antibody quantification | At baseline and on days 3, 7 and 21
Virology and immunological variables: Quantification of total antibodies in PC donors recovered from COVID-19. | Before infusion

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Hospital U. Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital U. Puerto Real, Puerto Real, Cádiz
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital U. Torrecárdenas, Almería
  - Hospital U. Puerta del Mar, Cadiz
  - Hospital U. Virgen de las Nieves, Granada
  - Hospital U. San Cecilio, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Regional U. de Málaga, Málaga
  - Hospital U. Virgen de la Victoria, Málaga
  - Hospital Unversitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital U. Nuestra Señora de Valme, Seville
  - Hospital San Juan de Dios, Seville